CLINICAL TRIAL: NCT01718119
Title: Phase III Clinical Trial Comparing the Efficacy and Safety of DA-3803(Recombinant Human Chorionic Gonadotrophin) and Ovidrel for Inducting Final Follicular Maturation and Early Luteinization in Women Undergoing Ovulation
Brief Title: Clinical Trial Comparing the Efficacy and Safety of DA-3803 and Ovidrel
Acronym: DA-3803
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA3803_HCG_III
Record Dates: First submitted 2012-02-05; First posted 2012-10-31 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Hyperovulation Induction for Assisted Reproduction Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DA-3803 (Experimental): subjects treated with DA-3803(r-hCG)
  Interventions: Drug: r-hCG
- Ovidrel (Active Comparator): subjects treated with Ovidrel(r-hCG)
  Interventions: Drug: r-hCG

INTERVENTIONS:
Drug: r-hCG — r-hCG(250mcg) injection subcutaneously

SUMMARY:
The purpose of this study is to compare the efficacy and safety of DA-3803(r-hCG) and Ovidrel for inducting final follicular maturation and early luteinization in women undergoing ovulation induction for assisted reproduction treatment

DETAILED DESCRIPTION:
This is an single-blind, randomized, comparative multicentric, phase III study to evaluate the safety and efficacy of DA-3803(r-hCG) in comparison with Ovidrel in the induction of final follicle maturation and early luteinization in 180 Korean female subjects undergoing superovulation. The study is organized on an outpatient basis in subjects undergoing assisted reproductive technologies (ART). The subjects are randomized into 2 groups. One group receive DA-3803(r-hCG) 250mcg and the other group receive Ovidrel®(r-hCG)250mcg. Each subject in both groups receives a single injection of hCG when the follicular development was judged to be adequate. Oocytes are retrieved 34-38 hours after r-hCG injection and fertilized in vitro. Not more than 4 embryos are to be replaced. Progesterone is administered daily according to center's normal practice, starting after the oocyte pick up and continuing until appropriate time. The subject is followed up and the treatment outcome (negative pregnancy test or pregnancy) is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Infertility regular ovulatory menstrual cycles : 25~35days
* BMI<=30kg/m2
* Early follicular phase serum levels are normal : FSH, LH, prolactin, testosterone
* Both ovaries present and clinically normal uterine cavity
* < 3 previous ART cycles, no ART cycles for 2 menstrual cycles
* semen analysis and ART are possible
* informed couple consent

Exclusion Criteria:

* With a poor response to gonadotrophin stimulation, such as ≤3 oocytes collected in any previous ART cycle
* Had previous severe ovarian hyperstimulation syndrome(OHSS)
* Polycystic ovarian syndrome(PCOS)
* Extra-uterine pregnancy within the last 3 months
* A clinically significant uncontrolled endocrine diseases, chronic cardiovascular disorders, hepatic, pulmonary and renal diseases
* Known allergy,hypersensitivity or contraindication to FSH, hCG, progesterone and GnRH antagonists
* medication with human gonadotrophin preparations(FSH, LH, hCG) within 2 months
* participation in another clinical trial within 1 month

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
the efficacy and safety of DA-3803(r-hCG) | about 1 month after ART
  the number of oocytes retrieved per patient following r-hCG administration, physical examination, clinical laboratory measurements, adverse events, injection-sited reactions, OHSS, number of multiple pregnancies

SECONDARY OUTCOMES:
the efficacy of DA-3803(r-hCG) | about 1 month after ART
  number of patients who received r-hCG with at least one oocyte retrieved, number of oocyte retrieved per number of follicles >10mm diameter on the day of r-hCG, number of mature oocytes, number of 2PN fertilized oocytes, number of 2PN cleaved embryos, implantation rate per embryo transferred, number of biochemical and clinical pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: TaeGi Yoon, MD, Study Chair — Cha Medical school Gangnam-Cha hospital; DongHee Choi, MD, Principal Investigator — Cha Medical school Boondang-Cha hospital; MiKyoung Goong, MD, Principal Investigator — Kwandong university medical school Cheil hospital
Locations (3):
- South Korea (3):
  - Cha Medical school Boondang-Cha hospital, Seongnam, Gyeong-Gi Do
  - Cha Medical school Gangnam-Cha hospital, Seoul
  - Kwandong university medical school Cheil hospital, Seoul